CLINICAL TRIAL: NCT00454935
Title: Correlation Between SV2A Expression in Tumour Tissue and Efficacy of Levetiracetam in Glioma Patients With Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Medical Center Haaglanden (Other)
Responsible Party: Prof Dr J.J. Heimans, VU University Medical Centre
Other Study IDs: EPI-GLIO-LEV
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Epilepsy; Glioma
Keywords: epilepsy; glioma
MeSH Terms: conditions — Epilepsy; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Tumor tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the correlation of SV2A expression in surgically removed tumour and tumour-surrounding tissue of glioma patients suffering from epilepsy with their clinical response to levetiracetam.

DETAILED DESCRIPTION:
Levetiracetam is a relatively novel anti-epileptic drug (AED), which has proven to be effective and well tolerated in many glioma patients with otherwise pharmacoresistant epilepsy. Moreover, levetiracetam has neither enzyme-inducing nor enzyme-inhibiting properties, which makes the drug particularly attractive for brain tumour patients, as they frequently receive chemotherapy and/or corticosteroids. Therefore, levetiracetam is the anti-epileptic drug of choice post-operatively in glioma patients suffering from epilepsy. Unfortunately, even with levetiracetam, a proportion of glioma patients is not free of seizures. It is unclear, however, which glioma patients benefit from levetiracetam treatment. It is suggested that the expression of protein SV2A is correlated with clinical response to levetiracetam. The determination of SV2A expression in brain (tumour) tissue might be used as a predictive tool for response to levetiracetam.

Objective of this study: Correlation of SV2A expression in surgically removed tumour and tumour-surrounding tissue of glioma patients suffering from epilepsy with their clinical response to levetiracetam.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* suffering from partial seizures, with or without secondary generalisation
* must have undergone surgery for their newly diagnosed or recurrent glioma not more than 42 days previously
* treated with levetiracetam
* histologically proven astrocytoma grade II or III, oligodendroglioma grade II or III, oligoastrocytoma grade II or III, or glioblastoma multiforme according to the World Health Organisation (WHO) classification of tumours affecting the central nervous system
* written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Patients who do not have a basic proficiency of the Dutch language,or are unable to communicate adequately will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult (> 18 years) glioma patients who suffer from partial seizures, with or without secondary generalisation, preoperatively. Patients must have undergone surgery for their newly diagnosed or recurrent glioma not more than 42 days previously and be treated with levetiracetam monotherapy at the time of inclusion.
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
to correlate the efficacy of post-operative levetiracetam monotherapy in newly diagnosed glioma patients suffering from epilepsy with expression of synaptic vesicle protein 2A (SV2A). | 6 months

SECONDARY OUTCOMES:
to determine the impact of levetiracetam monotherapy on neurocognitive functioning, health-related quality of life, and epileptic brain activity as measured by MEG, in newly diagnosed glioma patients with epilepsy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Heimans, prof. dr., Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Amsterdam, Netherlands